CLINICAL TRIAL: NCT00106275
Title: Mindfulness-Based Stress Reduction Program as an Intervention in Patients With Fibromyalgia: A Three-Armed Randomized Clinical Study
Brief Title: Mindfulness-Based Stress Reduction Program as an Intervention in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Samueli Institute for Information Biology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fibromyalgia & Mindfulness
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2005-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Meditation; Stress, Psychological; Monitoring, Ambulatory; Electrocardiographie, Ambulatory; Psychophysiology
MeSH Terms: conditions — Fibromyalgia; Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction

SUMMARY:
Fibromyalgia is a clinical syndrome with chronic pain, fatigue, and sleep disorders being the main symptoms. There is no commonly accepted efficacious treatment modality. Training in mindfulness-based stress reduction (MBSR) is a structured, 8-week, cognitively and affectively oriented intervention program, and has been shown to produce health benefits in a number of studies.

We plan to conduct a randomized, controlled, clinical study with the aim of testing the efficacy of MBSR for fibromyalgia. Because fibromyalgia is almost exclusively a female disorder, we will limit this investigation to women. 180 female, fibromyalgia patients will be randomized into three groups:

1. Mindfulness training
2. Active control
3. Wait-list control.

The main outcome criteria are self-reported and fibromyalgia-specific Quality of Life (QOL), and a Biobehavioral Fibromyalgia Index composed of a variety of psychophysiological and behavioral variables. This index will be generated from data gathered via an ambulatory psychophysiological monitoring system, which comprises parameters of mobility, sleep quality, and cardiovascular well-being. These and other relevant variables (depression score, general QOL, pain quality, anxiety, mindfulness, compliance, other therapeutic measures) will be assessed at the beginning and end of the training, as well as at 4- and 12-months post-treatment. A primary focus will be assessing whether it is possible to promote psychological well-being through the learning of attentive presence and any resultant affective affirmation.

DETAILED DESCRIPTION:
Background:

Fibromyalgia is a clinical syndrome with chronic pain, fatigue, and sleep disorders being the main symptoms. There is no commonly accepted efficacious treatment modality. Training in mindfulness meditation or mindfulness-based stress reduction(MBSR) is based on procedures derived from Buddhist insight meditation and developed into an eight-week structured program by Kabat-Zinn (e.g. 1982, Gen Hosp Psychiat 4:33-47). However, although mindfulness meditation derives from Buddhist practices, the procedures are completely nonesoteric and nonsectarian. In essence, it may be largely characterized in terms of a cognitively and affectively oriented intervention program, and has been shown to produce health benefits in a number of pilot studies, uncontrolled observational studies, and randomized investigations. Promising pilot data are also available for fibromyalgia patients. In a meta-analysis conducted by the PI (principal investigator), clinically important and statistically significant health benefits were found across individuals with a wide range of conditions.

Hypotheses:

1. A mindfulness-based stress reduction program (MBSR) is effective in improving the quality of life, psychological well-being and diminishing fibromyalgia-related symptoms in chronically ill patients;
2. the mindfulness component of the MBSR, a spiritual-based method, allows the patient to receive the energy of love which is then transformative; 3) the effects of the mindfulness training will be visible in physiologic measurements including autonomic nervous system activity.

Method and Results:

This is a randomized, controlled, clinical study with the aim of testing the efficacy of an MBSR for fibromyalgia. Because fibromyalgia is almost exclusively a female disorder, the investigation is limited to 180 female, fibromyalgia patients who will be randomized into three groups: Mindfulness training, Active control and Wait-list Control.

The main outcome criteria are self-reported and fibromyalgia-specific Quality of Life, and a Biobehavioral Fibromyalgia Index composed of a variety of psychophysiological and behavioral variables. This index will be generated from data parameters of mobility, sleep quality, and cardiovascular well-being. These and other relevant variables (depression score, general QOL, pain quality, anxiety, mindfulness, compliance, and other therapeutic measures) will be assessed at the beginning and end of the training, as well as at 4- and 12-months post-treatment. A primary focus will be assessing whether it is possible to promote psychological well-being through the learning of attentive presence and any resultant affective affirmation.

Anticipated Results:

MBSR will be proven to be a reliable and efficacious treatment for fibromyalgia as reflected in an improvement in patient reported health variables. It is also expected that a better understanding of the autonomic nervous system in the process of generating and maintaining fibromyalgia will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the German language
* Basic motivation to undergo a MBSR or similar training
* Motivation to participate in a clinical trial, especially to answer thoroughly the questionnaires
* Verified diagnosis of fibromyalgia according to the criteria of the American College of Rheumatology (ACR)

Exclusion Criteria:

* Life threatening disease
* Suppressed immune system
* Participation in other clinical trials
* Psychological or psychiatric disorders which constrain a normal interaction (assessed in an interview)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ)
Biobehavioral Fibromyalgia Index

SECONDARY OUTCOMES:
Quality of Life (PLC)
Pain sensation (SES)
Depression (ADS)
Anxiety (STAI-G)
Quality of sleep (SF-B)
Mindfulness (FIM)
Concomitant therapies
Compliance
Autonomic regulation
Physical activity measures
Sleep related measures

CONTACTS AND LOCATIONS:
Overall Officials: Paul Grossman, PhD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University Hospital Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Grossman P, Deuring G, Walach H, Schwarzer B, Schmidt S. Mindfulness-Based Intervention Does Not Influence Cardiac Autonomic Control or the Pattern of Physical Activity in Fibromyalgia During Daily Life: An Ambulatory, Multimeasure Randomized Controlled Trial. Clin J Pain. 2017 May;33(5):385-394. doi: 10.1097/AJP.0000000000000420. PMID 27518489
- See also: Study Description on the homepage of the funding institute — http://www.siib.org/Research_MandH_Schmidt2.asp